CLINICAL TRIAL: NCT06707584
Title: Role of MRI in Detection of Breast Cancer Molecular Subtypes in Correlation With Immunohistochemistry Results
Brief Title: Role of MRI in Breast Cancer Subtypes
Acronym: MRI
Status: Not yet recruiting | Type: Observational
Sponsor: Lamiaa Gomaa Ahmed Elsayed (Other)
Responsible Party: Sponsor-Investigator, Lamiaa Gomaa Ahmed Elsayed, Dr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MRI in breast cancer types
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: MRI in Breast Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
efficacy of MRI in detection of breast cancer molecular subtypes instead of biopsy and immunohistochemistry

DETAILED DESCRIPTION:
2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Patient with breast cancer (malignant breast mass) will do MRI breast and molecular subtypes will be assessed

MRI imaging studies will performed on a 1.5 T scanner , The patient is placed in the prone position with both breasts placed adequately in a double breast coil (four-channel phased array coil), MRI sequences are:

1. Axial T1WI. 2. Axial T2WI. 3. Axial STIR. 4. DCE-MRI with post-processing subtraction images 5- Axial DWI at b value( 0, 400, 800 and 1000 mm^2 per second) and ADC map will performed 6. MRI spectroscopy MRI acquisition protocol MRI protocols includes

* Axial T2-weighted fast spin echo sequence: TR=3840 ms, TE=81 ms, slice thickness=3.5 mm, and matrix=448×448.
* Coronal T2-weighted fast spin echo sequence: TR=3840 ms, TE=81 ms, slice thickness=3.5 mm, and matrix=448×448.s
* Short tau inversion recovery - axial: TR=8540 ms, TE=59 ms, TI=170 ms, slice thickness=3.5 mm, and matrix=320×314.4.
* The standard dynamic protocol commenced with a coronal three-dimensional rapid Field echo (thrive) sense non-enhanced T1-weighted sequence.
* A gadolinium containing contrast was administered at a dose of 0.2 ml/ kg by power injection at a speed of 2.0 ml/s and flushed with 20 ml of saline solution at the same rate.
* Dynamic imaging was then done in five consecutive series at 90-s intervals. Standard subtraction images were obtained by subtracting precontract images from the early peak postcontrast image.

ELIGIBILITY:
Inclusion Criteria:

a. patients with breast cancer confirmed by histopathology,

Exclusion Criteria:

1. breast implants
2. general Contraindication of MRI as claustrophobia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any patient with breast cancer
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-08-10 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of MRI in breast cancer subtyping | 5 years
  To investigate the diagnostic accuracy of dynamic post contrast imaging MRI in evaluation of breast cancer molecular subtypes and DWI and ADC in detection of breast cancer molecular subtypes